CLINICAL TRIAL: NCT05321745
Title: Repeated and Periodic Fecal Microbiota Transplantation in Children With Active and Refractory Crohn's Disease
Brief Title: Fecal Microbiota Transplantation in Pediatric Crohn's Disease
Acronym: FMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biao Zou (Other)
Responsible Party: Sponsor-Investigator, Biao Zou, attending physician, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20220127; TJ-IRB20220127 (Other: Tongji Hospital)
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Crohn Disease
Keywords: fecal microbiota transplantation , Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Partial enteral nutrition,FMT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repeated and multiple FMTs plus PEN (Experimental): repeated and multiple FMTs plus PEN(50% of total calories as polymeric diet, Peptamen, Nestle, Vevey, Switzerland) in refractory pediatric CD
  Interventions: Other: Standardized FMT

INTERVENTIONS:
Other: Standardized FMT — Fecal microbiota transplantation of fresh bacteria from healthy donor to the whole colon
  Other Names: Fecal Microbiota Transplantation

SUMMARY:
This study will test the safety and effectiveness of fecal microbiota transplantation (FMT) plus partial enteral nutrition (PEN) in refractory pediatric Crohn's disease (CD) who have failed conventional treatment

DETAILED DESCRIPTION:
Recent studies have suggested that gut imbalance and deregulation of immunological responses plays a pivotal role in the disease development of Crohn's disease (CD), and that FMT could be a useful treatment. Our study is aims to repeated and multiple FMTs plus PEN in the treatment of refractory pediatric CD. In the induction stage of CD, standard therapy remained unchanged, FMT and PEN were added, and FMT was given 1-2 courses, 3-6 times per course. In the maintaining stage, FMT was performed every 3 months, with the same 3-6 times of FMT treatment for each course, and the withdrawal of conventional drug therapy was gradually reduced. Refractory CD was defined as refractory to standard therapy (e.g., steroids, immunomodulators, cyclosporine, tacrolimus, or anti-TNF agents).

ELIGIBILITY:
Inclusion Criteria:

Aged 2-16 years and without genetic diseases; All refractory pediatric with mild-to-moderate CD; Mild-to-moderate CD, defined by the pediatric Crohn's disease activity index (PCDAI) >10 and ≤40 and Simple Endoscopic Score for CD (SES-CD) > 3 were enrolled in the study; refractory CD, defined by children who failed conventional treatment (hormone, immunosuppressant, biologics)

Exclusion Criteria Children who were treated by PEN (80%) less than 8 weeks; follow up less than 3 months; known contraindication to all FMT infusion method such as nasoduodenal tube insertion, oesophago-gastro-duodenoscopy (OGD), enteroscopy, colonoscopy, enema and Fecal capsule; unwilling to give informed consent/assent

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 8-12 weeks after FMT
  Clinical remission defined as a Pediatric Crohn's Disease Activity Index (PCDAI) score≤10
Endoscopic remission | 8-12 weeks after FMT
  Endoscopic remission defined by a Simple Endoscopic Score for CD （SES-CD) ≤ 2
Mucosal healing | 8-12 weeks after FMT
  Mucosal healing defined as SES-CD = 0

SECONDARY OUTCOMES:
Adverse events | 2 and 8 weeks after FMT
  All possible adverse events:fever,abdominal pain,infectious diseases and others

OTHER OUTCOMES:
gut microbial | before treatment and 4-8 weeks after treatment
  Fecal 16S RNA or macrogene sequencing was performed. Fecal samples were obtained from donor and recipient. The fecal samples and isolated microbiota samples were frozen immediately and underwent DNA extraction using standard methods.

CONTACTS AND LOCATIONS:
Overall Officials: Sainan Shu, MD, PhD, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zou B, Liu S, Dong C, Shen H, Lv Y, He J, Li X, Ruan M, Huang Z, Shu S. Fecal microbiota transplantation restores gut microbiota diversity in children with active Crohn's disease: a prospective trial. J Transl Med. 2025 Mar 6;23(1):288. doi: 10.1186/s12967-024-05832-1. PMID 40050917